CLINICAL TRIAL: NCT03595046
Title: The Evaluation of Erector Spinae Plane Block for the Pain Control of Thoracic Postherpetic Neuralgia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It was difficult to recruit subjects.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2018-0383
Record Dates: First submitted 2018-06-14; First posted 2018-07-23 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Thoracic Postherpetic Neuralgia
Keywords: thoracic paravertebral block; erector spinae plane block; thoracic postherpetic neuralgia
MeSH Terms: interventions — Ropivacaine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: erector spinae plane block group (group E) thoracic paravertebral block group (group P)
Who Masked: Participant, Investigator
Masking Description: 1. The subjects were randomly assigned to erector spinae plane block group (group E) and thoracic paravertebral block group (group P), and the assigned results are unknown.
  2. The Outcomes Assessor is not related to the study, and does not know its contents.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- erector spinae plane block group (group E) (Experimental): ultrasound-guided erector spinae plane block
  Interventions: Procedure: erector spinae plane block (20 mL of 0.25% ropivacaine with dexamethasone 5mg)
- thoracic paravertebral block group (group P) (Active Comparator): ultrasound-guided thoracic paravertebral block
  Interventions: Procedure: thoracic paravertebral block(10 mL 0.25% ropivacaine with dexamethasone 5mg)

INTERVENTIONS:
Procedure: erector spinae plane block (20 mL of 0.25% ropivacaine with dexamethasone 5mg) — In group E, The patient was placed in a sitting position and a high-frequency linear ultrasound transducer was placed in a longitudinal orientation 3 cm lateral to the thoracic spinous process. Three muscles were identified superficial to the hyperechoic transverse process shadow as follows: trapezius, rhomboid major, and erector spinae. An 8-cm 22-gauge block needle was inserted in a cephalad-to-caudad direction until the tip lay in the interfascial plane between transverse process and erector spinae muscles, as evidenced by visible linear spread of fluid between erector spinae muscles and the bony acoustic shadows of the transverse process. A total of 20 mL of 0.25% ropivacaine with dexamethasone 5mg was injected here.
  Arms: erector spinae plane block group (group E)
Procedure: thoracic paravertebral block(10 mL 0.25% ropivacaine with dexamethasone 5mg) — 2) In group P, an appropriate thoracic spinous precess is located by positioning the probe in the transverse plane. Then the probe is moved laterally to locate the transverse process. The probe is manipulated slightly caudad or cephala to locate the intercostal space. The transverse process is visualized medially with the pleura dipping under the inferolateral aspect. The internal intercostal membrane, which is contiguous with the superior costotransverse ligament, was generally seen as a thin, radiopaque line extending from the transverse process, creating a wedge-shaped pocket, which represents the thoracic paravertebral space. A 22-gauge, facet-tip needle is advanced, in plane, from the lateral aspect of the ultrasound probe. When the needle pierced the internal intercostal membrane, and after aspiration demonstrated the absence of air or blood, 10 mL 0.25% ropivacaine with dexamethasone 5mg deposited in 5-mL increments.
  Arms: thoracic paravertebral block group (group P)

SUMMARY:
Erector spinae plane block is new interfascial plane block, and can be applied to management of thoracic neuropathic pain syndromes. The target of needle is deeper(or anterior) to the erector spinae muscle. So it is more safe and simple technique than prior technique, thoracic paravertebral block. The aim of this study is the evaluation of erector spinae plane block comparison to prevertebra block.

DETAILED DESCRIPTION:
This study is single-blind because it is not possible to blind the practitioner performing the injection.

Subjects were randomly assigned to the erector spinae plane block group (group E) and the thoracic paravertebral block group (group P) by a random random number table, and the possibilities for belonging to any group were all the same and can not be artificially controlled by researchers.

Before the procedure, a resident who does not know of this study records the patient's pain and painDETECT. and on follow-up four weeks visits, PGIC scale is checked.

The erector spinae plane block or thoracic paravertebral block should be performed after receiving the informed consent of the patient.

Because of the large difference between the skilled and unskilled patients, the procedure in this study is performed by only one skilled practitioner.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria were patients who had chest wall post herpetic neuralgia, with moderate and severe pain and received appropriate antiviral therapy.

Exclusion Criteria:

1. Patient refusal
2. Patients who did not receive appropriate antiviral therapy
3. Patients with mild pain
4. Heavy skin eruption (no healthy area for needle entry) and infection at site of injection.
5. Patients with history of renal, hepatic diseases, coagulopathy, diabetes
6. Patients taking chemotherapy and/or radiotherapy
7. Patients with history of steroid therapy
8. Patients taking narcotic analgesics
9. Patient who does not understand the study because of illiteracy or language problems.
10. Abnormal findings in peripheral blood test (CBC, ESR, CRP, PT/aPTT)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-04-06 (Estimated); Study Completion 2019-06-06 (Estimated)

PRIMARY OUTCOMES:
1. Pain score (NRS) | Changes of Pain score from the procedure to 4 weeks
  1. in both groups, the patient is asked to score the pain before the procedure and 4 weeks later. And then the change of pain score is recorded.
  * NRS(numeric rating scale, on a scale of 0 to 10, with 0 being no pain at all and 10 being the worst pain imaginable)
2. painDETECT score | Changes of painDETECT score from the procedure to 4 weeks
  2. the patient is asked to painDETECT score the pain before the procedure and 4 weeks later. And then the change of painDETECT score is recorded.
  * painDETECT Questionnaire. The first five questions ask about the gradation of pain, scored from 0 to 5 (never = 0, hardly noticed = 1, slightly = 2; moderately = 3, strongly = 4, very strongly = 5). Question 6 asks about the pain course pattern, scored from -1 to 2, depending on which pain course pattern diagram is selected. Question 7 asks about radiating pain, answered as yes or no, and scored as 2 or 0 respectively. The total score summed each subscales is between -1 and 38, indicates the likelihood of a neuropathic pain component. A score less than 12 indicates that pain is unlikely to have a neuropathic component, while a score more than 19 suggests that pain is likely to have a neuropathic component.
3. PGIC, 7 scales(overall improvement of pain relief) | Changes of PGIC, 7 scales from the procedure to 4 weeks
  3. the patient is asked to PGIC, 7 scales about overall improvement of pain relief 4 weeks later.
  * Patient's global impression of change(PGIC) scale. Since beginning treatment at this clinic, the change (if any) in ACTIVITY LIMITATIONS, SYMPTOMS, EMOTIONS, and OVERALL QUALITY OF LIFE, related to your painful condition. (No change =1, almost the same = 2, a little better = 3, somewhat better =4, moderate better =5, better =6, a great deal better =7)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No